CLINICAL TRIAL: NCT03524612
Title: A Phase II, Open-label, Prospective, Single-arm, Study to Assess Ability of Eltrombopag to Induce Sustained Remission in Subjects With ITP Who Are Refractory or Relapsed After First-line Steroids
Brief Title: A Study to Assess the Ability of Eltrombopag to Induce Sustained Response Off Treatment in Subjects With ITP
Acronym: TAPER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CETB115J2411; 2018-000452-18 (EudraCT Number)
Record Dates: First submitted 2018-05-02; First posted 2018-05-15 (Actual); Results first posted 2023-12-27 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Immune Thrombocytopenic Purpura (ITP)
Keywords: Thrombocytopenic; Immune; Platelets; Bleeding; ITP; eltrombopag; ETB115; induce sustained response off treatment; refractory or relapsed; first-line steroids
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Hemorrhage; Recurrence | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- eltrombopag (Other): Participants were treated with eltrombopag to induce sustained response off treatment to reach a target platelet count of >=100×10^9/L (CR), after 1st line steroids had failed.
  Interventions: Drug: eltrombopag

INTERVENTIONS:
Drug: eltrombopag — 12.5, 25, 50 and 75 mg tablets for oral use once daily
  Other Names: ETB115

SUMMARY:
The purpose of this trial was to assess the ability of eltrombopag to induce sustained treatment-free remission in immune thrombocytopenia purpura (ITP) subjects who relapsed or failed to respond to an initial treatment with steroids.

DETAILED DESCRIPTION:
Protocol Amendment 01 added a follow-up period of 12 months for patients with sustained response off treatment at month 12 to obtain further data on response duration.

The starting dose was eltrombopag 50 mg daily (25 mg daily for Asian patients and 12.5 mg daily for Japanese patients in Japan). The starting dose for this study was consistent with the dosing guidelines approved for eltrombopag use in ITP. An increase of eltrombopag dose up to 75 mg was allowed for patients who did not respond to standard-dosage treatment and to reduce the risk of bleeding. The rationale for this increased dose was to use the minimal efficacious dosage of eltrombopag in order to achieve a platelet count ≥ 100×10^9/L and maintain it around 100×10^9/L (no counts below 70×10^9/L) for 2 months in order to allow patients to start the eltrombopag tapering and withdrawal process.

Patients who reached a platelet count of >= 100 × 10^9/L and maintained counts around 100×10^9/L for 2 months with no platelet count < 70 × 10^9/L were eligible for tapering-off and treatment discontinuation, which occurred via 25 mg reduction every 2 weeks up to 25 mg on alternate days for 2 weeks until treatment discontinuation.

Patients who successfully discontinue eltrombopag and maintained platelet count >= 30 × 10^9/L in the absence of bleeding or use of rescue therapy were followed to month 12. If a relapse (defined as platelet count <30 × 10^9/L) occurred during the 12-month treatment period, they were offered a new course of eltrombopag treatment within this timeframe at the appropriate starting dose. If a patient relapsed in the post 12-month follow-up period, no further attempts for tapering and achieving sustained response off treatment were made.

The taper-off scheme followed recommendations within the current established dosing regimen for when to consider dose adjustment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained prior to participation in the study
2. Patients ≥ 18 years old
3. Patients with a confirmed diagnosis of primary ITP, who are not responsive or in relapse after a first line of steroid therapy ± intravenous immunoglobulin (IVIG) (used as a rescue therapy)
4. Platelet count < 30×10^9/L and assessed as needing treatment (per physician's discretion

Exclusion Criteria:

1. ITP patients previously treated with any ITP second-line therapies, thrombopoietin receptor (TPO-R) agonists for ITP, except steroids / IVIG
2. Patients who relapsed more than one year after the end of first-line full course of steroid therapy
3. Patients with a diagnosis of secondary thrombocytopenia
4. Patients who have life threatening bleeding complications per investigator discretion
5. Patients who had a deep vein thrombosis or arterial thrombosis in the 6 months preceding enrollment
6. Serum creatinine ≥ 1.5 mg/dL
7. Total bilirubin > 1.5 × upper limit of normal (ULN)
8. Aspartate transaminase (AST) > 3.0 × ULN
9. Alanine transaminase (ALT) > 3.0 × ULN
10. Patients who are human immune deficiency virus (HIV), hepatitis C virus (HCV), hepatitis B surface antigen (HBsAg) positive
11. Patients with hepatic impairment (Child-Pugh score > 5)
12. Patients who have active malignancy
13. Patients with any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions that could interfere with subject's safety, obtaining informed consent or compliance with the study procedures per investigator discretion
14. History or current diagnosis of cardiac disease indicating significant risk of safety for Patients participating in the study
15. Patients with known active or uncontrolled infections not responding to appropriate therapy
16. Patients with evidence of current alcohol/drug abuse
17. Women of child-bearing potential and sexually active males unwilling to use adequate contraception during the study
18. Female Patients who are nursing or pregnant (positive serum or urine B-human chorionic gonadotrophin (B-hCG) pregnancy test) at screening or pre-dose on Day 1

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2022-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (30):
- United States (2):
  - Hematology Oncology Association of Rockland, Nyack, New York
  - Case Western Reserve, Cleveland, Ohio
- Novartis Investigative Site, Linz, Austria
- Brazil (3):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, São Paulo, São Paulo
- Chile (2):
  - Novartis Investigative Site, Temuco, Región de la Araucanía
  - Novartis Investigative Site, Viña del Mar, Región de Valparaíso
- France (2):
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Pessac
- Greece (2):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Pátrai
- Italy (2):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Trieste, TS
- Novartis Investigative Site, Nagoya, Aichi-ken, Japan
- Mexico (2):
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Mexico City
- Novartis Investigative Site, Muscat, Oman
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Spain (5):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Murcia
- Novartis Investigative Site, Bern, Switzerland
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Aydin
  - Novartis Investigative Site, Edirne
  - Novartis Investigative Site, Kocaeli
- Novartis Investigative Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Cooper N, Ghanima W, Vianelli N, Valcarcel D, Yavasoglu I, Melikyan A, Ruiz EY, Haenig J, Somenzi O, Lee J, Clark J, Zhang Y, Zaja F. Sustained response off-treatment in eltrombopag-treated adult patients with ITP who are refractory or relapsed after first-line steroids: Primary, final, and ad-hoc analyses of the Phase II TAPER trial. Am J Hematol. 2024 Jan;99(1):57-67. doi: 10.1002/ajh.27131. Epub 2023 Nov 28. PMID 38014779

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 32 investigative sites in 15 countries:1 (Austria), 3 (Brazil), 2 (Chile), 2 (France), 2 (Greece), 2 (Italy), 1 (Japan), 2 (Mexico), 1 (Oman), 2 (Russia), 7 (Spain), 1 (Switzerland), 3 (Turkey), 1 (UK), 2 (USA).
Period: Overall Study
Arm/Group | Eltrombopag
Started (All patients were included in the Full Analysis Set (FAS) and Safety Set (SAF)) | 105
Completed | 63
Not Completed | 42
Not completed — Lack of Efficacy | 10
Not completed — Physician Decision (Patient non-compliant) | 1
Not completed — Adverse Event | 10
Not completed — Withdrawal by Subject | 7
Not completed — Patient Decision (Patient Changed Her Address) | 1
Not completed — Patient Decision (Personal Reasons) | 1
Not completed — New therapy for study indication | 6
Not completed — Death | 3
Not completed — Lost to Follow-up | 2
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Eltrombopag
Number analyzed (Participants) | 105
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.1 (19.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 95
  More than one race | 0
  Unknown or Not Reported | 1
Time since initial diagnosis [Mean (Standard Deviation); unit: Days] — Time since initial diagnosis is the difference in days between the date of initial diagnosis and the date of first dose of eltrombopag.
  Days | 366.37 (911.420)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Response Off Treatment (SRoT) by 12 Months
Description: Sustained response off treatment (SRoT) was defined as: reaching platelet count >= 100×10^9/L (complete response [CR]) and then maintaining platelet counts around 100×10^9/L for 2 months (no counts below 70×10^9/L), AND then tapering off the drug until treatment discontinuation while maintaining platelet count >= 30×10^9/L in the absence of bleeding (no bleeding AEs) or use of any rescue therapy until month 12.
Time Frame: Month 12
Population: Full Analysis Set, which included all patients who received at least one dose of eltrombopag.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 105
Percentage of participants | 30.5 [21.9 to 40.2]
Statistical Analysis 1: Comparison: Eltrombopag; Test type: Other; p < 0.0001, Clopper Pearson test

2. Secondary Outcome: Median Duration of Sustained Response Off Treatment (SRoT) After Treatment Discontinuation for Participants With Sustained Response Off Treatment
Description: as for outcome 1
Time Frame: From last dose of eltrombopag to month 12
Population: Full Analysis Set
Measure: Median (Full Range); unit: Weeks
Arm/Group | Eltrombopag
Number analyzed (Participants) | 105
Weeks | 33.3 [4 to 51]

3. Secondary Outcome: Estimated Median Duration of Sustained Response Off Treatment (SRoT) for Participants With Sustained Response Off Treatment at Month 12 and Who Enter 12 Months Follow-up Period
Description: Sustained response off treatment (SRoT) was defined as: reaching platelet count >= 100×10^9/L (complete response [CR]) and then maintaining platelet counts around 100×10^9/L for 2 months (no counts below 70×10^9/L), AND then tapering off the drug until treatment discontinuation while maintaining platelet count >= 30×10^9/L in the absence of bleeding (no bleeding AEs) or use of any rescue therapy.
  Patients with SRoT until month 12 who entered follow-up and did not relapse by cut-off date/Month 24 were censored at the earliest of discontinuation date/death date/Month 24 platelet assessment date/cutoff date. Patients with SRoT until Month 12 patients who did not enter or do not yet have data in follow-up phase are censored at their Month 12 platelet assessment date.
Time Frame: From last dose of eltrombopag to relapse, assessed up to month 24
Population: Full Analysis Set. No data collected for this endpoint.
Arm/Group | Eltrombopag
Number analyzed (Participants) | 0

4. Secondary Outcome: Estimated Median Duration of Sustained Response Off Treatment (SRot) for All Patients
Description: Patients who tapered and discontinued successfully, or did not relapse/die by cutoff date /month 24 were censored at the earliest of discontinuation date/death date/month 24 platelet assessment date/cutoff date.
Time Frame: From last dose of eltrombopag to month 24
Population: Full Analysis Set. No data collected for this endpoint.
Arm/Group | Eltrombopag
Number analyzed (Participants) | 0

5. Secondary Outcome: Percentage of Participants With Sustained Response Off Treatment Until Month 24
Description: Sustained response off treatment is defined as reach platelet count ≥ 100×10^9/L (complete response [CR]) and then maintain platelet counts around 100×10^9/L for 2 months (no counts below 70×10^9/L) AND then taper off the drug until treatment discontinuation while, maintain platelet count ≥ 30×10^9/L in the absence of bleeding (no bleeding AEs) or use of any rescue therapy
Time Frame: Month 15, 18, 21 and 24
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 105
Participants
  Month 15 | 21
  Month 18 | 18
  Month 21 | 14
  Month 24 | 15

6. Secondary Outcome: Percentage of Participants With Early Response Within First Month
Description: Early response is defined as reaching a platelet count >= 50×10^9/L at least once within the first month (month 1) without bleeding events and no rescue therapy.
Time Frame: By 1 month
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 105
Percentage of participants | 76.2 [66.9 to 84.0]

7. Secondary Outcome: Percentage of Participants With Recovery Response in Case of Loss of Response During or After Tapering of Eltrombopag Until Month 24
Description: Recovery response is defined as platelet count >=30×10^9/L after eltrombopag is re-introduced, in case of loss of response (< 30×10^9/L and/or bleeding event) without bleeding events and no rescue therapy.
Time Frame: Up to month 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 105
Percentage of participants
  Participants with loss of response | 11.4 [6.0 to 19.1]
  Participants with recovery response | 6.7 [2.7 to 13.3]

8. Secondary Outcome: Relative Change From Baseline in Platelet Count Over Time
Description: Relative change (%) is the absolute change divided by the platelet counts at baseline and multiplied by 100.
Time Frame: Baseline, month 3, 6, 9, 12 (End of Treatment Visit for non-responders), 15, 18, 21 and 24 (End of Treatment Visit for responders), assessed up to 12 months for non-responders and up to 24 months for responders
Population: Full Analysis Set. Only participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Eltrombopag
Number analyzed (Participants) | 104
Percentage of change
  3 Months: number analyzed (Participants) | 86
  3 Months | 1384.29 (3383.702)
  6 Months: number analyzed (Participants) | 72
  6 Months | 1313.10 (3459.616)
  9 Months: number analyzed (Participants) | 66
  9 Months | 1396.68 (3238.680)
  12 Months: number analyzed (Participants) | 69
  12 Months | 1464.95 (3509.964)
  15 Months: number analyzed (Participants) | 35
  15 Months | 1622.19 (3712.156)
  18 Months: number analyzed (Participants) | 30
  18 Months | 1664.90 (3718.191)
  21 Months: number analyzed (Participants) | 28
  21 Months | 2527.20 (5098.612)
  24 Months: number analyzed (Participants) | 28
  24 Months | 1691.68 (3611.977)
  end of treatment visit | 1213.91 (2952.719)

9. Secondary Outcome: Percentage of Participants Who Maintain Platelet Counts Level Within 12 Months and Every 3 Months Until Month 24
Description: Platelet counts level is defined as having platelet counts >=30×10^9/L without bleeding events and no rescue therapy.
Time Frame: From first time of reaching the level to month 3, 6, 9, 12 (End of Treatment Visit for non-responders), 15, 18, 21 and 24 (End of Treatment Visit for responders), assessed up to 12 months for non-responders and up to 24 months for responders
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 105
Percentage of participants
  maintain platelet counts level from the first time of reaching that level to month 3 | 49.5 [39.6 to 59.5]
  maintain platelet counts level from the first time of reaching that level to month 6 | 38.1 [28.8 to 48.1]
  maintain platelet counts level from the first time of reaching that level to month 9 | 28.6 [20.2 to 38.2]
  maintain platelet counts level from the first time of reaching that level to month 12 | 28.6 [20.2 to 38.2]
  maintain platelet counts level from the first time of reaching that level to month 15 | 20.0 [12.8 to 28.9]
  maintain platelet counts level from the first time of reaching that level to month 18 | 17.1 [10.5 to 25.7]
  maintain platelet counts level from the first time of reaching that level to month 21 | 13.3 [7.5 to 21.4]
  maintain platelet counts level from the first time of reaching that level to month 24 | 14.3 [8.2 to 22.5]
  maintain platelet counts level from the first time of reaching that level to end of treatment visit | 31.4 [22.7 to 41.2]

10. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Questionaire
Description: The Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue©) is a 13- item questionnaire that assesses self-reported fatigue and its impact upon daily activities over the past 7 days. FACIT-fatigue is scored using a 4-point Likert scale. Items are scored as follows: 4 = Not At All; 3 = A Little Bit; 2 = Somewhat; 1 = Quite A Bit; 0 = Very Much, EXCEPT items #7 and #8 which are reversed scored. Score range from 0-52. A score of less than 30 indicates severe fatigue. The higher the score, the better the quality of life (less fatigue).
Time Frame: Baseline to month 3, 6, 9, 12 (End of Treatment Visit for non-responders), 15, 18, 21 and 24 (End of Treatment Visit for responders), assessed up to 12 months for non-responders and up to 24 months for responders
Population: Full Analysis Set. Only participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Eltrombopag
Number analyzed (Participants) | 85
Unit on a scale
  3 Months: number analyzed (Participants) | 66
  3 Months | 5.42 (9.700)
  6 Months: number analyzed (Participants) | 62
  6 Months | 6.15 (8.779)
  9 Months: number analyzed (Participants) | 45
  9 Months | 6.89 (9.291)
  12 Months: number analyzed (Participants) | 58
  12 Months | 7.90 (9.064)
  15 Months: number analyzed (Participants) | 25
  15 Months | 7.12 (11.720)
  18 Months: number analyzed (Participants) | 23
  18 Months | 8.87 (11.644)
  21 Months: number analyzed (Participants) | 22
  21 Months | 8.80 (11.112)
  24 Months: number analyzed (Participants) | 26
  24 Months | 8.69 (10.635)
  end of treatment visit | 5.40 (10.116)

11. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy- Thrombocytopenia (FACT-Th6) Questionnaire
Description: FACT-Th6 instrument is used to measure worry/concern about bleeding and bruising, and the impact of this worry/concern on physical and social activity (Cella 2006). FACT-Th6 is a 6-item subset of the more detailed FACT-Th, which is an 18-item subscale of the validated FACT that specifically measures concerns related to thrombocytopenia in the past 7 days. The FACT-Th6 is scored using a 5-level Likert scale (0=not at all to 4=very much) and is calculated by summing scores for the 6-items; therefore, scores can range from 0-24, with higher scores representing better HRQoL
Time Frame: as for outcome 10
Population: Full Analysis Set. Only participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Eltrombopag
Number analyzed (Participants) | 85
Unit on a scale
  3 Months: number analyzed (Participants) | 66
  3 Months | 3.80 (5.130)
  6 Months: number analyzed (Participants) | 62
  6 Months | 4.35 (6.312)
  9 Months: number analyzed (Participants) | 45
  9 Months | 5.60 (6.114)
  12 Months: number analyzed (Participants) | 58
  12 Months | 5.62 (6.505)
  15 Months: number analyzed (Participants) | 25
  15 Months | 5.44 (8.949)
  18 Months: number analyzed (Participants) | 23
  18 Months | 7.04 (7.654)
  21 Months: number analyzed (Participants) | 22
  21 Months | 7.32 (7.351)
  24 Months: number analyzed (Participants) | 26
  24 Months | 7.08 (7.048)
  end of treatment visit | 4.15 (6.631)

12. Secondary Outcome: Change From Baseline in Short Form 36 Health Survey (SF-36v2) Questionnaire: Bodily Pain (BP) Score
Description: The SF-36 Scale is a 36-item, patient-reported survey which measures overall quality of life. It consists of 8 subscales (bodily pain (BP), general health (GH), mental health (MH), physical functioning (PF), role emotional (SE), role physical (RP), social role functioning (SF) and vitality (VT)) which can be aggregated to derive a physical-component summary (PCS) score and a mental-component score (MCS). The SF-36 is scored using norm-based scoring procedures: each sub-scale score ranges from 0 to 10, and the composite score ranges from 0 to 100. Higher scores indicative of better HRQoL.
Time Frame: as for outcome 10
Population: Full Analysis Set. Only participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Eltrombopag
Number analyzed (Participants) | 85
Unit on a scale
  3 Months: number analyzed (Participants) | 66
  3 Months | 7.55 (24.199)
  6 Months: number analyzed (Participants) | 61
  6 Months | 2.75 (24.636)
  9 Months: number analyzed (Participants) | 45
  9 Months | 3.82 (21.507)
  12 Months: number analyzed (Participants) | 58
  12 Months | 7.53 (25.547)
  15 Months: number analyzed (Participants) | 24
  15 Months | 1.96 (36.697)
  18 Months: number analyzed (Participants) | 23
  18 Months | 13.61 (26.662)
  21 Months: number analyzed (Participants) | 22
  21 Months | 3.00 (20.967)
  24 Months: number analyzed (Participants) | 26
  24 Months | 9.27 (29.090)
  end of treatment visit | 5.19 (29.460)

13. Secondary Outcome: Change From Baseline in Short Form 36 Health Survey (SF-36v2) Questionnaire: General Health (GH) Score
Description: as for outcome 12
Time Frame: as for outcome 10
Population: Full Analysis Set. Only participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Eltrombopag
Number analyzed (Participants) | 85
Unit on a scale
  3 Months: number analyzed (Participants) | 66
  3 Months | 4.12 (18.894)
  6 Months: number analyzed (Participants) | 61
  6 Months | 5.39 (20.646)
  9 Months: number analyzed (Participants) | 45
  9 Months | 7.40 (17.990)
  12 Months: number analyzed (Participants) | 58
  12 Months | 7.62 (18.420)
  15 Months: number analyzed (Participants) | 24
  15 Months | 11.17 (20.470)
  18 Months: number analyzed (Participants) | 23
  18 Months | 14.78 (26.801)
  21 Months: number analyzed (Participants) | 22
  21 Months | 14.36 (25.541)
  24 Months: number analyzed (Participants) | 26
  24 Months | 13.92 (19.577)
  end of treatment visit | 3.80 (18.122)

14. Secondary Outcome: Change From Baseline in Short Form 36 Health Survey (SF-36v2) Questionnaire: Mental Health (MH) Score
Description: as for outcome 12
Time Frame: as for outcome 10
Population: Full Analysis Set. Only participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Eltrombopag
Number analyzed (Participants) | 85
Unit on a scale
  3 Months: number analyzed (Participants) | 66
  3 Months | 6.74 (15.775)
  6 Months: number analyzed (Participants) | 61
  6 Months | 6.97 (18.149)
  9 Months: number analyzed (Participants) | 45
  9 Months | 9.78 (15.074)
  12 Months: number analyzed (Participants) | 58
  12 Months | 10.26 (16.125)
  15 Months: number analyzed (Participants) | 24
  15 Months | 7.08 (22.259)
  18 Months: number analyzed (Participants) | 23
  18 Months | 15.22 (22.334)
  21 Months: number analyzed (Participants) | 22
  21 Months | 14.32 (20.948)
  24 Months: number analyzed (Participants) | 26
  24 Months | 12.50 (17.103)
  end of treatment visit | 6.82 (17.058)

15. Secondary Outcome: Change From Baseline in Short Form 36 Health Survey (SF-36v2) Questionnaire: Physical Functioning (PF) Score
Description: as for outcome 12
Time Frame: as for outcome 10
Population: Full Analysis Set. Only participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Eltrombopag
Number analyzed (Participants) | 85
Unit on a scale
  3 Months: number analyzed (Participants) | 66
  3 Months | 8.48 (23.842)
  6 Months: number analyzed (Participants) | 61
  6 Months | 10.90 (26.069)
  9 Months: number analyzed (Participants) | 45
  9 Months | 12.67 (28.074)
  12 Months: number analyzed (Participants) | 58
  12 Months | 14.31 (28.767)
  15 Months: number analyzed (Participants) | 24
  15 Months | 11.87 (37.469)
  18 Months: number analyzed (Participants) | 23
  18 Months | 19.35 (33.449)
  21 Months: number analyzed (Participants) | 22
  21 Months | 24.09 (31.983)
  24 Months: number analyzed (Participants) | 26
  24 Months | 16.54 (35.882)
  end of treatment visit | 9.00 (29.376)

16. Secondary Outcome: Change From Baseline in Short Form 36 Health Survey (SF-36v2) Questionnaire: Role Emotional (RE) Score
Description: as for outcome 12
Time Frame: as for outcome 10
Population: Full Analysis Set. Only participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Eltrombopag
Number analyzed (Participants) | 85
Unit on a scale
  3 Months: number analyzed (Participants) | 66
  3 Months | 4.42 (22.371)
  6 Months: number analyzed (Participants) | 61
  6 Months | 6.15 (23.270)
  9 Months: number analyzed (Participants) | 45
  9 Months | 8.89 (22.361)
  12 Months: number analyzed (Participants) | 58
  12 Months | 10.20 (23.260)
  15 Months: number analyzed (Participants) | 24
  15 Months | 4.86 (27.022)
  18 Months: number analyzed (Participants) | 23
  18 Months | 13.04 (26.211)
  21 Months: number analyzed (Participants) | 22
  21 Months | 16.29 (25.520)
  24 Months: number analyzed (Participants) | 26
  24 Months | 16.03 (20.128)
  end of treatment visit | 7.25 (22.078)

17. Secondary Outcome: Change From Baseline in Short Form 36 Health Survey (SF-36v2) Questionnaire: Role Physical (RP) Score
Description: as for outcome 12
Time Frame: as for outcome 10
Population: Full Analysis Set. Only participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Eltrombopag
Number analyzed (Participants) | 85
Unit on a scale
  3 Months: number analyzed (Participants) | 66
  3 Months | 13.26 (22.958)
  6 Months: number analyzed (Participants) | 61
  6 Months | 9.43 (27.066)
  9 Months: number analyzed (Participants) | 45
  9 Months | 17.36 (24.165)
  12 Months: number analyzed (Participants) | 58
  12 Months | 19.94 (29.232)
  15 Months: number analyzed (Participants) | 24
  15 Months | 15.89 (37.454)
  18 Months: number analyzed (Participants) | 23
  18 Months | 22.55 (32.680)
  21 Months: number analyzed (Participants) | 22
  21 Months | 27.27 (33.604)
  24 Months: number analyzed (Participants) | 26
  24 Months | 29.81 (32.849)
  end of treatment visit | 15.88 (33.332)

18. Secondary Outcome: Change From Baseline in Short Form 36 Health Survey (SF-36v2) Questionnaire: Social Functioning (SF) Score
Description: as for outcome 12
Time Frame: as for outcome 10
Population: Full Analysis Set. Only participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Eltrombopag
Number analyzed (Participants) | 85
Unit on a scale
  3 Months: number analyzed (Participants) | 66
  3 Months | 6.06 (24.143)
  6 Months: number analyzed (Participants) | 61
  6 Months | 7.17 (26.951)
  9 Months: number analyzed (Participants) | 45
  9 Months | 10.00 (22.863)
  12 Months: number analyzed (Participants) | 58
  12 Months | 16.38 (26.408)
  15 Months: number analyzed (Participants) | 24
  15 Months | 14.58 (30.986)
  18 Months: number analyzed (Participants) | 23
  18 Months | 26.63 (24.514)
  21 Months: number analyzed (Participants) | 22
  21 Months | 20.45 (26.318)
  24 Months: number analyzed (Participants) | 26
  24 Months | 25.96 (22.617)
  end of treatment visit | 11.18 (26.236)

19. Secondary Outcome: Change From Baseline in Short Form 36 Health Survey (SF-36v2) Questionnaire: Vitality (VT) Score
Description: as for outcome 12
Time Frame: as for outcome 10
Population: Full Analysis Set. Only participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Eltrombopag
Number analyzed (Participants) | 85
Unit on a scale
  3 Months: number analyzed (Participants) | 66
  3 Months | 7.48 (18.418)
  6 Months: number analyzed (Participants) | 61
  6 Months | 6.45 (20.696)
  9 Months: number analyzed (Participants) | 45
  9 Months | 12.78 (20.982)
  12 Months: number analyzed (Participants) | 58
  12 Months | 14.33 (22.398)
  15 Months: number analyzed (Participants) | 24
  15 Months | 8.33 (26.237)
  18 Months: number analyzed (Participants) | 23
  18 Months | 12.23 (27.918)
  21 Months: number analyzed (Participants) | 22
  21 Months | 17.33 (26.087)
  24 Months: number analyzed (Participants) | 26
  24 Months | 11.06 (24.705)
  end of treatment visit | 8.97 (22.503)

20. Secondary Outcome: Change From Baseline in Short Form 36 Health Survey (SF-36v2) Questionnaire: Physical Component Summary (PCS) Score
Description: as for outcome 12
Time Frame: as for outcome 10
Population: Full Analysis Set. Only participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Eltrombopag
Number analyzed (Participants) | 85
Unit on a scale
  3 Months: number analyzed (Participants) | 66
  3 Months | 3.46 (7.445)
  6 Months: number analyzed (Participants) | 61
  6 Months | 2.72 (8.165)
  9 Months: number analyzed (Participants) | 45
  9 Months | 3.92 (7.608)
  12 Months: number analyzed (Participants) | 58
  12 Months | 4.85 (8.946)
  15 Months: number analyzed (Participants) | 24
  15 Months | 4.37 (11.754)
  18 Months: number analyzed (Participants) | 23
  18 Months | 6.77 (9.950)
  21 Months: number analyzed (Participants) | 22
  21 Months | 6.65 (8.017)
  24 Months: number analyzed (Participants) | 26
  24 Months | 6.63 (9.627)
  end of treatment visit | 3.30 (9.728)

21. Secondary Outcome: Change From Baseline in Short Form 36 Health Survey (SF-36v2) Questionnaire: Mental Component Summary (MCS) Score
Description: as for outcome 12
Time Frame: as for outcome 10
Population: Full Analysis Set. Only participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Eltrombopag
Number analyzed (Participants) | 85
Unit on a scale
  3 Months: number analyzed (Participants) | 66
  3 Months | 2.34 (8.443)
  6 Months: number analyzed (Participants) | 61
  6 Months | 2.85 (9.451)
  9 Months: number analyzed (Participants) | 45
  9 Months | 4.52 (7.815)
  12 Months: number analyzed (Participants) | 58
  12 Months | 5.33 (8.719)
  15 Months: number analyzed (Participants) | 24
  15 Months | 3.28 (11.083)
  18 Months: number analyzed (Participants) | 23
  18 Months | 7.12 (11.312)
  21 Months: number analyzed (Participants) | 22
  21 Months | 7.18 (11.143)
  24 Months: number analyzed (Participants) | 26
  24 Months | 6.87 (9.081)
  end of treatment visit | 3.53 (9.002)

22. Secondary Outcome: Percentage of Participants With Worst Post-baseline Value in Functional Assessment of Cancer Therapy-G (GP5)
Description: The GP5 is a single question used to assess the overall bothersomeness of treatment side effects. The GP5 is scored using a 5-point rating scale (0 = not at all; 1 = a little bit; 2 = somewhat; 3 = quite a bit; and 4 = very much), where lower scores reflect less bothersomeness from treatment side effects.
Time Frame: Baseline to end of treatment visit, assessed up to 12 months for non-responders and up to 24 months for responders
Population: Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 105
Participants
  Rating 0 | 51
  Rating 1 | 15
  Rating 2 | 10
  Rating 3 | 2
  Rating 4 | 5
  Missing | 22

23. Secondary Outcome: Overall Change of Treatment Satisfaction Using Treatment Satisfaction Questionnaire (TSQM-9)
Description: The Treatment Satisfaction Questionnaire for Medication (TSQM-9) is a psychometric measure of a patient's satisfaction with medication. It consists of 3 subscales: effectiveness, convenience and global satisfaction. The scores were computed by adding items for each domain, i.e. 1 to 3 for effectiveness, 4 - 6 for convenience and 7 to 9 for global satisfaction. The lowest possible score (1 for each item and 3 for all 3 subscales) was subtracted from the composite score and divided by the greatest possible score range. The greatest range was (7-1) X 3 items = 18 for the effectiveness and convenience, and (5-1) x 3 items = 12 for global satisfaction. This provided a transformed score between 0 and 1 that was then multiplied by 100. A positive change from baseline indicates improvement.
Time Frame: Baseline to month 12 (End of Treatment Visit for non-responders) and 24 (End of Treatment Visit for responders), assessed up to 12 months for non-responders and up to 24 months for responders
Population: Full Analysis Set. Only participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Eltrombopag
Number analyzed (Participants) | 66
Unit on a scale
  Global Satisfaction change from BL at 12 months: number analyzed (Participants) | 49
  Global Satisfaction change from BL at 12 months | 17.78 (29.201)
  Global Satisfaction change from BL at 24 months: number analyzed (Participants) | 21
  Global Satisfaction change from BL at 24 months | 17.69 (26.110)
  Global Satisfaction change from BL at end of treatment visit | 9.96 (33.966)
  Effectiveness change from BL at 12 months: number analyzed (Participants) | 49
  Effectiveness change from BL at 12 months | 18.82 (33.809)
  Effectiveness change from BL at 24 months: number analyzed (Participants) | 21
  Effectiveness change from BL at 24 months | 17.99 (29.913)
  Effectiveness change from BL at end of treatment visit | 14.14 (36.673)
  Convenience change from BL at 12 months: number analyzed (Participants) | 49
  Convenience change from BL at 12 months | 17.69 (30.758)
  Convenience change from BL at 24 months: number analyzed (Participants) | 21
  Convenience change from BL at 24 months | 19.05 (25.189)
  Convenience change from BL at end of treatment visit | 15.07 (30.253)
  Total score change from BL at 12 months: number analyzed (Participants) | 49
  Total score change from BL at 12 months | 54.29 (78.218)
  Total score change from BL at 24 months: number analyzed (Participants) | 21
  Total score change from BL at 24 months | 54.72 (75.463)
  Total score change from BL at end of treatment visit | 39.17 (86.449)

24. Post Hoc Outcome: All Collected Deaths
Description: On-treatment deaths were reported from the date of first dose of eltrombopag to 30 days after the date of the last non-zero dose of eltrombopag for patients who discontinued on or before month 12 (i.e., non-responders). For patients ongoing at month 12, the on-treatment period lasted until the cut-off date for the primary analysis (22-Oct-2021; approximately 35 months), as a patient could restart treatment at any time during study.
  Post-treatment deaths were collected in the post treatment period from 31 days after last dose of study medication until the cut-off date for the primary analysis (22-Oct-2021; approximately 35 months). These are not considered Adverse Events.
Time Frame: On-treatment deaths: Up to approximately 35 months. Post-treatment deaths: Up to approximately 35 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 105
Participants
  On-treatment deaths | 3
  Post-treatment deaths: number analyzed (Participants) | 102
  Post-treatment deaths | 1
  All deaths | 4

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days for patients who discontinued on or before month 12. For patients ongoing at month 12, the on-treatment period lasted until the cut-off date for the primary analysis (22-Oct-2021), up to a maximum of 35 months).Deaths were collected in the post treatment follow up period from 31 days after last dose of study medication until the cut-off date for the primary analysis (22-Oct-2021).
Description: Any sign or symptom that occurred during the conduct of the trial and safety follow-up.
Groups:
- Eltrombopag (On-Treatment): Participants were treated with eltrombopag to induce sustained response off treatment to reach a target platelet count of >=100×10^9/L (CR), after 1st line steroids had failed.
- Eltrombopag (Post-treatment Follow-up): Deaths collected in the post- treatment follow-up period (starting from day 31 post- treatment). No AEs were collected during this period.
Arm/Group | Eltrombopag (On-Treatment) | Eltrombopag (Post-treatment Follow-up)
All-Cause Mortality (participants affected / at risk) | 3/105 | 1/102
Serious Adverse Events (participants affected / at risk) | 21/105 | 0/0
Other Adverse Events (participants affected / at risk) | 64/105 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (On-Treatment) (N=105) | Eltrombopag (Post-treatment Follow-up) (N=0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | NA
Diarrhoea (Gastrointestinal disorders) | 1 | NA
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | NA
Vomiting (Gastrointestinal disorders) | 1 | NA
Cholecystitis acute (Hepatobiliary disorders) | 1 | NA
Cavernous sinus thrombosis (Infections and infestations) | 1 | NA
Diarrhoea infectious (Infections and infestations) | 1 | NA
Peritonsillar abscess (Infections and infestations) | 1 | NA
Tuberculosis (Infections and infestations) | 1 | NA
Intentional product misuse (Injury, poisoning and procedural complications) | 2 | NA
Platelet count decreased (Investigations) | 2 | NA
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | NA
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | NA
Carotid artery stenosis (Nervous system disorders) | 1 | NA
Central nervous system haemorrhage (Nervous system disorders) | 1 | NA
Cerebral haemorrhage (Nervous system disorders) | 1 | NA
Haemorrhage intracranial (Nervous system disorders) | 1 | NA
Acute kidney injury (Renal and urinary disorders) | 1 | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Petechiae (Skin and subcutaneous tissue disorders) | 1 | NA
Deep vein thrombosis (Vascular disorders) | 1 | NA
Superficial vein thrombosis (Vascular disorders) | 1 | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (On-Treatment) (N=105) | Eltrombopag (Post-treatment Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 7 | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 16 | NA
Abdominal pain (Gastrointestinal disorders) | 7 | NA
Diarrhoea (Gastrointestinal disorders) | 10 | NA
Gingival bleeding (Gastrointestinal disorders) | 6 | NA
Nausea (Gastrointestinal disorders) | 8 | NA
Vomiting (Gastrointestinal disorders) | 6 | NA
Asthenia (General disorders) | 8 | NA
Fatigue (General disorders) | 6 | NA
Alanine aminotransferase increased (Investigations) | 9 | NA
Aspartate aminotransferase increased (Investigations) | 6 | NA
Blood alkaline phosphatase increased (Investigations) | 7 | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | NA
Headache (Nervous system disorders) | 23 | NA
Petechiae (Skin and subcutaneous tissue disorders) | 11 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/12/NCT03524612/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-07): https://cdn.clinicaltrials.gov/large-docs/12/NCT03524612/SAP_001.pdf